CLINICAL TRIAL: NCT06827782
Title: Clinical Study of Cord Blood-derived CAR-NK Cells Targeting CD19 in the Treatment of Refractory/Relapsed Central Nervous System Lymphoma
Brief Title: Cord Blood-derived CAR-NK Cells Targeting CD19 for Refractory/Relapsed Central Nervous System Lymphoma
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID2024482
Record Dates: First submitted 2024-12-29; First posted 2025-02-14 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2024-12

CONDITIONS: Refractory/Recurrent Central Nervous System Lymphoma
Keywords: Refractory or recurrent; central nervous system lymphoma; Diffuse large B cell lymphoma; CAR-NK
MeSH Terms: conditions — Recurrence; Lymphoma, Large B-Cell, Diffuse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CB CAR-NK019 (Experimental)
  Interventions: Biological: anti-CD19 CAR-NK cells

INTERVENTIONS:
Biological: anti-CD19 CAR-NK cells — lentiviral vector-transducted cord blood-derived NK cells to express anti-CD19 CAR

SUMMARY:
This study is designed to evaluate the safety and efficacy of cord blood-derived CAR-NK019 in the treatment of refractory/relapsed central nervous system lymphoma.

DETAILED DESCRIPTION:
This study is a single-center, open, single-arm incremental, exploratory study designed to evaluate the safety and efficacy of cord blood-derived CAR-NK019 in the treatment of refractory/relapsed central nervous system lymphoma.

The study will be divided into two stages: Phase I is the dose escalation study, which is strictly based on the "3+3" dose escalation principle, and three dose groups are set up, which are administered through the ommaya capsule ventricle, and each dose is infused once a week for 3 weeks. Three to six subjects are intended to be enrolled in each dose group, with each subject observed for at least 28 days after receiving the initial infusion and a long-term follow-up period of two years after each infusion. Phase II is the dose expansion phase: The recommended dose and administration mode for this phase will be determined after comprehensive consideration based on safety data obtained in phase I, the proliferation and survival of CAR-NK cells in vivo, and clinical efficacy data, and 24 effective subjects will be recruited for further evaluation of efficacy and safety. Long-term follow-up lasted up to 2 years after the first CAR-NK transfusion in each patient.

ELIGIBILITY:
Inclusion Criteria:

* Patients with refractory/recurrent CNS lymphoma must meet all of the following criteria to be eligible:

  1. Voluntarily participate in the study and sign the informed consent;
  2. Age 18-75 years old, male or female;
  3. Diffuse large B-cell lymphoma (DLBCL) was confirmed by histology. CD19 expression was positive by lymphoma pathology or flow cytometry, and CD19 expression was ≥20% by IHC.
  4. Imaging showed no evidence of systemic lymphoma;
  5. Meets any of the following definitions for refractory/relapsed CNS lymphoma: no complete response has been achieved with prior 2-line regimen including methotrexate or cytarabine-based regimen; Disease progression during any treatment; The stable time of disease after effective treatment is less than 6 months; Disease progression or recurrence within 12 months after autologous hematopoietic stem cell transplantation.
  6. Imaging showed the presence of at least one measurable lesion, with a minimum diameter of ≥10mm;
  7. Expected survival ≥3 months;
  8. ECOG score 0-3 points;
  9. Adequate organ function reserve:

     * alanine aminotransferase, ASpartate aminotransferase ≤ 2.5× UNL (upper limit of normal);
     * Creatinine clearance (Cockcroft-Gault method) ≥60 mL/min;
     * Serum total bilirubin and alkaline phosphatase ≤1.5× UNL;
     * Glomerular filtration rate >50ml/min
     * cardiac ejection fraction (EF) ≥45%;
     * Basic oxygen saturation >92% in indoor natural air environment;
     * Blood routine: absolute number of neutrophils >×109/L, platelet count 45×109/L, hemoglobin 80g/L;
  10. Previous autologous hematopoietic stem cell transplantation is allowed, and the interval between stem cell transfusion and CAR-NK transfusion is ≥3 months;
  11. Previous CAR-T cell therapy is allowed, and the time interval between CAR-T transfusion and CAR-NK transfusion is ≥3 months;
  12. Female subjects of childbearing age must test negative for pregnancy and agree to use effective contraception during the test;
  13. Approved anti-tumor therapies, such as systemic chemotherapy, whole body radiotherapy and immunotherapy, have been discontinued for at least 3 weeks before the study; Discontinuation of targeted drug regiments without chemotherapy for at least 2 weeks;

Exclusion Criteria:

* Subjects who meet any of the following criteria will not be admitted to the study:

  1. Allergic to any of the components of cell products;
  2. History of other tumors;
  3. Acute grade II-IV (Glucksberg standard) GvHD or generalized chronic GvHD occurred after previous allogeneic hematopoietic stem cell transplantation; Or are receiving anti-GVHD treatment;
  4. Have received gene therapy within the past 3 months;
  5. Active infections requiring treatment (except simple urinary tract infections, bacterial pharyngitis), but prophylactic antibiotic, antiviral and antifungal infection treatment is permitted;
  6. Persons infected with hepatitis B (HBsAg positive, but HBV-DNA<103 is not excluded) or hepatitis C virus (including virus carriers), syphilis and other acquired and congenital immunodeficiency diseases, including but not limited to HIV-infected persons;
  7. Subjects with Grade III or IV cardiac dysfunction according to the New York Heart Association's cardiac function grading criteria;
  8. Patients who received antitumor therapy in the early stage but did not recover toxicity (CTCAE 5.0 toxicity did not recover to ≤ grade 1, except fatigue, anorexia, alopecia);
  9. Previous history of epilepsy, autoimmune encephalitis, cerebral infarction or cerebral hemorrhage within 6 months;
  10. Whole-body enhanced CT or PET/CT suggests evidence of systemic lymphoma;
  11. Lactating women who are unwilling to stop breastfeeding;
  12. Any other circumstances that the investigator believes may increase the risk to the subject or interfere with the test results;
  13. Patients requiring more than 10mg of dexamethasone per day for 3 days prior to enrollment;
  14. Patients who cannot tolerate ommaya capsule implantation;
  15. Those who cannot tolerate enhanced magnetic resonance imaging.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2025-03-01 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicity (DLTs) | Up to 28 days
  To evaluate the safety, tolerability, and determine the recommended dosage of cord blood-derived Anti-CD19 CAR-NK Cell Therapy for refractory/relapsed central nervous system lymphoma

SECONDARY OUTCOMES:
Complete response rate (CR) | 3 months
  To determine the anti-tumor effectivity of CB CAR-NK019
Overall response rate (ORR) | 3 months
  To determine the anti-tumor effectivity of CB CAR-NK019
Progression free survival (PFS) | Up to 2 years
  To determine the anti-tumor effectivity of CB CAR-NK019
Overall survival (OS) | Up to 2 years
  To determine the anti-tumor effectivity of CB CAR-NK019
Duration of response (DOR) | Up to 2 years
  To determine the anti-tumor effectivity of CB CAR-NK019

CONTACTS AND LOCATIONS:
Locations (1):
- 2nd Affiliated Hospital, School of Medicine, Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No